CLINICAL TRIAL: NCT04026672
Title: Hemp Oil + User Experience Study: A Retrospective, Non-Interventional Study to Assess Consumer Experience and the Impact of Hemp Oil + on Quality of Life
Brief Title: Hemp Oil + User Experience Study
Status: Completed | Type: Observational
Sponsor: Thorne HealthTech, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: Hemp-PM001
Record Dates: First submitted 2019-06-28; First posted 2019-07-19 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: General Wellbeing; Gastrointestinal Health; Physical Discomfort; Sleep; Mood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Presented as an online survey, this study seeks to better understand how Thorne customers are using and experiencing the new Hemp Oil + product and how they feel it compares in the marketplace. Hemp Oil + is a combination product with a proprietary blend of hemp, clove, black pepper, hops, and rosemary extracts. People who have independently elected to purchase and use Hemp Oil + before the study starts will be invited to voluntarily participate. If they meet study requirements and give consent they will answer questions online about their experience with Hemp Oil +. Questions address general demographics and wellness, general impressions of the product, how it compares to other products, and any effect it has had on their gastrointestinal health, physical discomfort, sleep, and mood. The survey is expected to take 15-30 min of participant time. Data will be analyzed to determine whether the customer experience with Hemp Oil + is as favorable as it seems from anecdotal reports. Analysis will also be conducted to find patterns that can inform future studies, marketing, and customer education efforts.

ELIGIBILITY:
Inclusion Criteria:

* Has personally used at least one bottle (30 gelcaps) of Hemp Oil +
* Provides consent to participate in the study

Exclusion Criteria:

* Cannot access or use the electronic survey for any reason
* Was pregnant or nursing when taking Hemp Oil +
* Is a Thorne employee not willing to participate without compensation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People who have purchased Hemp Oil +
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Assess impact to overall quality of life (QoL) after taking Hemp Oil + | 1 Day
  Questionnaire gathering data from the past 30 or more days

SECONDARY OUTCOMES:
Assess impact to specific QoL factors - GI health, mood, sleep, physical discomfort - after taking Hemp Oil + | 1 Day
  Questionnaire gathering data from the past 30 or more days
Gain insight into user perspective on product quality, efficacy, and rationale for continuing/discontinuing use | 1 Day
  Questionnaire gathering data from the past 30 or more days

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Jacques, ND, Principal Investigator — Thorne Research; Sheena Smith, MS, Principal Investigator — Thorne Research
Locations (1):
- Online Survey for Thorne Research, Inc., Summerville, South Carolina, United States